CLINICAL TRIAL: NCT01613794
Title: Prospective Randomized Controlled, Open Label, Clinical Trial to Study if Rosuvastatin Use Improves the Coagulation Profile in Patients With Venous Thrombosis
Brief Title: Rosuvastatin Use to Improve the Coagulation Profile in Patients With Venous Thrombosis
Acronym: START
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Leiden University Medical Center (Other)
Collaborators: Netherlands Heart Foundation (Other)
Responsible Party: Principal Investigator, Willem M. Lijfering, Principal Investigator, Leiden University Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 2011T012; 2012-000223-41 (EudraCT Number)
Record Dates: First submitted 2012-05-31; First posted 2012-06-07 (Estimated); Last update posted 2017-01-16 (Estimated); Status verified 2017-01

CONDITIONS: Deep Vein Thrombosis; Pulmonary Embolism
Keywords: Deep vein thrombosis; Pulmonary embolism; Rosuvastatin treatment; Pharmacologic actions
MeSH Terms: conditions — Venous Thrombosis; Pulmonary Embolism | interventions — Rosuvastatin Calcium

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- No intervention (No Intervention)
- Rosuvastatin (Experimental)
  Interventions: Drug: Rosuvastatin

INTERVENTIONS:
Drug: Rosuvastatin — 20 mg od
  Other Names: crestor
  Arms: Rosuvastatin

SUMMARY:
Epidemiological studies have shown a 2-3 fold increased long-term risk of arterial cardiovascular disease after venous thrombosis, most predominant in the first year following initial venous thrombosis. The results of recent observational studies that showed 40-50% risk reductions for first venous thrombosis occurrence when using a statin are in this aspect promising. The results are also somewhat surprising, because the mechanism behind this effect is unclear. Dyslipidemia may be the most plausible explanation to be considered. However, as dyslipidemia is not related to an increased risk of venous thrombosis, it is unlikely that statins decrease venous thrombosis risk by lipid lowering activities. Recent observations indicate that coagulation can activate the initial formation of atherosclerosis. Our hypothesis is therefore that the coagulation profile in persons with venous thrombosis is improved when using a statin, ultimately leading to less atherosclerosis: another well known property of statin use.

ELIGIBILITY:
Inclusion Criteria:

* Provision of informed consent prior to any study specific procedures
* Persons with (initial or recurrent) confirmed symptomatic proximal deep vein thrombosis or pulmonary embolism who after a time period of at least 3 to 12 months are allowed to stop, - or stopped using < 1 month anticoagulant treatment as indicated by their treating physician
* Persons aged 18 years or above

Exclusion Criteria:

* Persons already using statins or lipid lowering drugs, or any other disallowed concomitant medications (erythromycin, HIV protease inhibitors, or cyclosporine)
* History of statin-induced myopathy, or serious hypersensitivity reaction to other HMG-CoA reductase inhibitors (statins), including rosuvastatin
* Life expectancy less than 6 months
* Pregnant woman or woman with childbearing potential who are not willing to use contraception
* Active liver or kidney disease or dysfunction or muscle disorders
* Unstable medical or psychological condition that interferes with study participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 255 (Actual)
Dates: Start 2012-12; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Coagulation factor VIII | 28 days
  Change in factor VIII level from baseline to 28 days of intervention

CONTACTS AND LOCATIONS:
Locations (3):
- Netherlands (3):
  - Trombosedienst Medial, Hoofddorp, South Holland
  - Leiden anticoagulation clinic, Leiden, South Holland
  - Erasmus Medical Center, Rotterdam

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Lijfering WM, Flinterman LE, Vandenbroucke JP, Rosendaal FR, Cannegieter SC. Relationship between venous and arterial thrombosis: a review of the literature from a causal perspective. Semin Thromb Hemost. 2011 Nov;37(8):885-96. doi: 10.1055/s-0031-1297367. Epub 2011 Dec 23. PMID 22198853
- [Derived] Ramberg C, Hindberg K, Biedermann JS, Cannegieter SC, van der Meer FJ, Snir O, Leebeek FWG, Kruip MJHA, Hansen JB, Lijfering WM. Rosuvastatin treatment decreases plasma procoagulant phospholipid activity after a VTE: A randomized controlled trial. J Thromb Haemost. 2022 Apr;20(4):877-887. doi: 10.1111/jth.15626. Epub 2022 Jan 8. PMID 34953155
- [Derived] Biedermann JS, Cannegieter SC, Roest M, van der Meer FJ, Reitsma PH, Kruip MJ, Lijfering WM. Platelet reactivity in patients with venous thrombosis who use rosuvastatin: a randomized controlled clinical trial. J Thromb Haemost. 2016 Jul;14(7):1404-9. doi: 10.1111/jth.13343. Epub 2016 Jun 10. PMID 27094802
- [Derived] Lippi G, Favaloro EJ, Sanchis-Gomar F. Venous thrombosis associated with HMG-CoA reductase inhibitors. Semin Thromb Hemost. 2013 Jul;39(5):515-32. doi: 10.1055/s-0033-1343892. Epub 2013 Apr 29. PMID 23629822